CLINICAL TRIAL: NCT00093730
Title: Phase I Study Of BMS-599626 In Patients With Advanced Solid Malignancies That Express Her2
Brief Title: BMS-599626 in Treating Patients With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000389510; UCLA-0404066-01; BMS-CA181002
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

ARMS (1):
- BMS-59926 (Experimental)
  Interventions: Drug: BMS-59926

INTERVENTIONS:
Drug: BMS-59926

SUMMARY:
RATIONALE: BMS-599626 may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase I trial is studying the side effects and best dose of BMS-599626 in treating patients with metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose, biologically active dose, and recommended phase II dose(s) of BMS-599626 in patients with metastatic HER2/neu-overexpressing primary solid tumors.

Secondary

* Determine the safety and tolerability of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the effect of this drug on biomarkers and predictive markers of HER1 and HER2 in skin and tumor in these patients.
* Evaluate tumor metabolic activity in response to this drug in these patients.
* Determine, preliminarily, evidence of anti-tumor activity of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive oral BMS-599626 once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BMS-599626 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 20 patients are treated at that dose level.

PROJECTED ACCRUAL: Approximately 3-60 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary solid (i.e., non-hematologic) tumor

  * Radiographic or tissue confirmation of metastatic disease

    * Locally advanced disease allowed if no surgical or local therapeutic treatment exists
* HER2/neu overexpression (1+, 2+, or 3 +) by immunohistochemistry

  * Tumors with HER2 gene amplification by fluorescence in situ hybridization analysis allowed
* Tumor paraffin tissue block OR 20-30 unstained slides from tumor tissue block must be available for biomarker and predictive marker analyses
* Disease progression during or after standard therapy OR no standard therapy exists
* Measurable or non-measurable disease

  * Measurable disease is required for the expanded cohort treated at the maximum tolerated dose of the study drug
* No known brain metastasis

  * Patients with controlled brain metastasis with no disease progression 60 days after prior therapy and no neurologic signs or symptoms are allowed

    * Patients with signs or symptoms suggestive of brain metastasis are eligible provided that brain metastasis is ruled out by CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN
* PT/PTT ≤ 1.5 times ULN
* INR ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN
* Calcium normal

Cardiovascular

* LVEF ≥ 45%
* Heart rate ≥ 50 beats/min on electrocardiogram
* No uncontrolled cardiovascular disease
* No myocardial infarction within the past 12 months
* No uncontrolled angina within the past 6 months
* No congestive heart failure within the past 6 months
* No prolonged QTc (> 450 msec) on electrocardiogram
* No diagnosed or suspected congenital long QT syndrome
* No history of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
* No history of second- or third-degree heart block

  * Patients with pacemakers may be eligible
* No uncontrolled hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study participation
* Potassium normal
* Magnesium normal
* No medical condition that has a risk of causing torsades de pointes
* No active infection
* No serious uncontrolled medical disorder that would preclude study participation
* No dementia or altered mental status that would preclude giving informed consent
* No known allergy to BMS-599626 or related compound
* No prisoners or patients involuntarily incarcerated for treatment of either a psychiatric or physical (e.g., infectious disease) illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior immunotherapy
* At least 2 weeks since prior targeted kinase inhibitor (e.g., trastuzumab [Herceptin^®])

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, or doxorubicin HCl liposome)

Endocrine therapy

* At least 2 weeks since prior anticancer hormonal therapy

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* Recovered from prior therapy
* Prior adjuvant or neoadjuvant therapy allowed
* No short-acting antacids (e.g., Maalox^® or TUMS^®) 8 hours before or 4 hours after study drug administration
* No recent anticancer therapy
* More than 4 weeks since prior investigational agents
* At least 5 days (or 5 half-lives) since prior drugs that cause torsades de pointes
* At least 48 hours since prior proton pump inhibitors (e.g., omeprazole or lansoprazole) or histamine H_2 antagonists (e.g., ranitidine, famotidine, or cimetidine)
* Concurrent low-dose coumadin allowed
* No other concurrent investigational agents
* No concurrent drugs that may cause torsades de pointes or QTc prolongation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-08; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose of BMS-599626 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Pegram, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States